CLINICAL TRIAL: NCT06589258
Title: Study of the Passage of (CBD) Into Breast Milk and Its Biological Impact on Breast-fed Children
Brief Title: Cannabidiol Into Breastmilk
Acronym: CBD-ALLT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUO-2024-02
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Breast Feeding
Keywords: cannabidiol; Breast milk; Breast-feeding; Breast-feed children; PK POP
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: One group of sixty breastfeeding mothers with CBD's consumption
  Two subgroups: thirty subjects by group:
  * only CBD intake
  * CBD and others psychoactive substances
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- breastfeeding mothers with CBD's consumption (Other): Determination of delta 9-tetrahydrocannabinol (THC) and its metabolites , and of cannabidiol and its metabolites in blood and breast-milk by liquid chromatography-tandem mass spectrometry (LC-MS/MS). Realization of THC/CBD ratio; qualitative research in mother's and breast-fed child's urine for the presence of cannabinoids (THC, CBD and its metabolites).
  Interventions: Biological: Assessing maternal and lactational plasma CBD uptake at different stages of breastfeeding

INTERVENTIONS:
Biological: Assessing maternal and lactational plasma CBD uptake at different stages of breastfeeding — Determination of delta 9-tetrahydrocannabinol (THC) and its metabolites , and of cannabidiol and its metabolites in blood and breasts-milk by liquid chromatography-tandem mass spectrometry (LC-MS/MS). Realization of THC/CBD ratio; qualitative research in mother's and breast-fed child's urine for the presence of cannabinoids (THC, CBD and its metabolites).

SUMMARY:
Really few data published to date on the passage of CBD into breast milk. The investigators known that 17.5 percent of the French human being between 18 and 34 years old consume CBD and among this, nearly half are women. None official French data to say how many French breastfeeding mothers consume CBD. CBD is a legal, psychoactive but not psychoaddictive substance. CBD's pharmacokinetic and pharmacodynamics make us fear that CBD could easily go through mother's milk. No published data available on possible effect in breast-fed child, not even on possible biological passage in breast-fed child. The aim of his study is to evaluate the passage of CBD in blood and milk at different moments of the breastfeeding (mothers) and its possible found in the infants'urine.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18
* Breastfeeding CBD user
* Having given written informed consent

Exclusion Criteria:

* Women who do not understand French well
* Women with a psychiatric or dual pathology that prevents proper participation in the study,
* Women under protective supervision (guardianship/curatorship),
* Women under court protection,
* Women not affiliated to a social security scheme

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Theoretical dose of CBD received by the breastfed child over 24 hours | Day 2 postpartum
  Theoretical dose of CBD received by the breastfed child over 24 hours by measuring blood and milk concentrations of CBD during postpartum visits.
Theoretical dose of CBD received by the breastfed child over 24 hours | Day 21 postpartum
  Theoretical dose of CBD received by the breastfed child over 24 hours by measuring blood and milk concentrations of CBD during postpartum visits.
Theoretical dose of CBD received by the breastfed child over 24 hours | Day 42 postpartum
  Theoretical dose of CBD received by the breastfed child over 24 hours by measuring blood and milk concentrations of CBD during postpartum visits.
Theoretical dose of CBD received by the breastfed child over 24 hours | Month 3 postpartum
  Theoretical dose of CBD received by the breastfed child over 24 hours by measuring blood and milk concentrations of CBD during postpartum visits.
Theoretical dose of CBD received by the breastfed child over 24 hours | Month 4 postpartum
  Theoretical dose of CBD received by the breastfed child over 24 hours by measuring blood and milk concentrations of CBD during postpartum visits.
Theoretical dose of CBD received by the breastfed child over 24 hours | Month 6 postpartum
  Theoretical dose of CBD received by the breastfed child over 24 hours by measuring blood and milk concentrations of CBD during postpartum visits.
Theoretical dose of CBD received by the breastfed child over 24 hours | Month 9 postpartum
  Theoretical dose of CBD received by the breastfed child over 24 hours by measuring blood and milk concentrations of CBD during postpartum visits.
Theoretical dose of CBD received by the breastfed child over 24 hours | Month 12 postpartum
  Theoretical dose of CBD received by the breastfed child over 24 hours by measuring blood and milk concentrations of CBD during postpartum visits.

SECONDARY OUTCOMES:
Concentration of CBD in maternal blood | Day 2 postpartum
Concentration of CBD in maternal blood | Day 21 postpartum
Concentration of CBD in maternal blood | Day 42 postpartum
Concentration of CBD in maternal blood | Month 3 postpartum
Concentration of CBD in maternal blood | Month 4 postpartum
Concentration of CBD in maternal blood | Month 6 postpartum
Concentration of CBD in maternal blood | Month 9 postpartum
Concentration of CBD in maternal blood | Month 12 postpartum
Concentration of CBD metabolites in maternal blood | Day 2 postpartum
Concentration of CBD metabolites in maternal blood | Day 21 postpartum
Concentration of CBD metabolites in maternal blood | Month 3 postpartum
Concentration of CBD metabolites in maternal blood | Month 4 postpartum
Concentration of CBD metabolites in maternal blood | Month 6 postpartum
Concentration of CBD metabolites in maternal blood | Month 9 postpartum
Concentration of CBD metabolites in maternal blood | Month 12 postpartum
Concentration of CBD in breast-milk | Day 2 postpartum
Concentration of CBD in breast-milk | Day 21 postpartum
Concentration of CBD in breast-milk | Day 42 postpartum
Concentration of CBD in breast-milk | Month 3 postpartum
Concentration of CBD in breast-milk | Month 4 postpartum
Concentration of CBD in breast-milk | Month 6 postpartum
Concentration of CBD in breast-milk | Month 9 postpartum
Concentration of CBD in breast-milk | Month 12 postpartum
THC concentrations in mother's blood | Day 2 postpartum
THC concentrations in mother's blood | Day 21 postpartum
THC concentrations in mother's blood | Day 42 postpartum
THC concentrations in mother's blood | Month 3 postpartum
THC concentrations in mother's blood | Month 4 postpartum
THC concentrations in mother's blood | Month 6 postpartum
THC concentrations in mother's blood | Month 9 postpartum
THC concentrations in mother's blood | Month 12 postpartum
THC concentrations in breast milk | Day 2 postpartum
THC concentrations in breast milk | Day 21 postpartum
THC concentrations in breast milk | Day 42 postpartum
THC concentrations in breast milk | Month 3 postpartum
THC concentrations in breast milk | Month 4 postpartum
THC concentrations in breast milk | Month 6 postpartum
THC concentrations in breast milk | Month 9 postpartum
THC concentrations in breast milk | Month 12 postpartum
Percentage of breastfeeding mother's with CBD metabolites in urine | Day 2 postpartum
Percentage of breastfeeding mother's with CBD metabolites in urine | Day 21 postpartum
Percentage of breastfeeding mother's with CBD metabolites in urine | Day 42 postpartum
Percentage of breastfeeding mother's with CBD metabolites in urine | Month 3 postpartum
Percentage of breastfeeding mother's with CBD metabolites in urine | Month 4 postpartum
Percentage of breastfeeding mother's with CBD metabolites in urine | Month 6 postpartum
Percentage of breastfeeding mother's with CBD metabolites in urine | Month 9 postpartum
THC/CBD ratio | Day 2 postpartum
Percentage of breastfeeding child with CBD in urine | Day 2 postpartum
Percentage of breastfeeding child with CBD in urine | Day 21 postpartum
Percentage of breastfeeding child with CBD in urine | Day 42 postpartum
Percentage of breastfeeding child with CBD in urine | Month 3 postpartum
Percentage of breastfeeding child with CBD in urine | Month 4 postpartum
Percentage of breastfeeding child with CBD in urine | Month 6 postpartum
Percentage of breastfeeding child with CBD in urine | Month 9 postpartum
Percentage of breastfeeding child with CBD metabolites in urine | Day 2 postpartum
Percentage of breastfeeding child with CBD metabolites in urine | Day 21 postpartum
Percentage of breastfeeding child with CBD metabolites in urine | Day 42 postpartum
Percentage of breastfeeding child with CBD metabolites in urine | Month 3 postpartum
Percentage of breastfeeding child with CBD metabolites in urine | Month 4 postpartum
Percentage of breastfeeding child with CBD metabolites in urine | Month 6 postpartum
Percentage of breastfeeding child with CBD metabolites in urine | Month 9 postpartum
impact of ethnicity | Day 2 postpartum
Percentage of breastfeeding mother's with CBD in urine | Day 2 postpartum
Percentage of breastfeeding mother's with CBD in urine | Day 21 postpartum
Percentage of breastfeeding mother's with CBD in urine | Day 42 postpartum
Percentage of breastfeeding mother's with CBD in urine | Month 4 postpartum
Percentage of breastfeeding mother's with CBD in urine | Month 6 postpartum
Percentage of breastfeeding mother's with CBD metabolites in urine | Month 12 postpartum
Percentage of breastfeeding mother's with CBD in urine | Month 12 postpartum
Percentage of breastfeeding mother's with CBD in urine | Month 3 postpartum
Percentage of breastfeeding child with CBD metabolites in urine | Month 12 postpartum
Percentage of breastfeeding mother's with THC in urine | Day 2 postpartum
Percentage of breastfeeding mother's with THC in urine | Day 21 postpartum
Percentage of breastfeeding mother's with THC in urine | Day 42 postpartum
Percentage of breastfeeding mother's with THC in urine | Month 3 postpartum
Percentage of breastfeeding mother's with THC in urine | Month 4 postpartum
Percentage of breastfeeding mother's with THC in urine | Month 6 postpartum
Percentage of breastfeeding mother's with THC in urine | Month 9 postpartum
Percentage of breastfeeding mother's with THC in urine | Month 12 postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Philippe LEBOUCHARD-MAAKAROUN, Dr, Principal Investigator — CHU Orleans
Locations (1):
- CHU Orléans, Orléans, France

REFERENCES:
- [Background] Kessler FH, von Diemen L, Ornell F, Sordi AO. Cannabidiol and mental health: possibilities, uncertainties, and controversies for addiction treatment. Braz J Psychiatry. 2021 Sep-Oct;43(5):455-457. doi: 10.1590/1516-4446-2021-1838. No abstract available. PMID 34008796
- [Background] Costentin J. [Epigenetic effects of cannabis/tetrahydrocannabinol]. Bull Acad Natl Med. 2020 Jun;204(6):570-576. doi: 10.1016/j.banm.2020.04.004. Epub 2020 Apr 15. French. PMID 32296244
- [Background] Potenza MN, Bunt G, Khalsa JH. Addiction Medicine Physicians and Medicinal Cannabinoids. JAMA Psychiatry. 2023 Jul 1;80(7):659-660. doi: 10.1001/jamapsychiatry.2023.0731. PMID 37133830
- [Background] Johnson CT, Bradshaw HB. Modulatory Potential of Cannabidiol on the Opioid-Induced Inflammatory Response. Cannabis Cannabinoid Res. 2021 Jun;6(3):211-220. doi: 10.1089/can.2020.0181. PMID 34115948
- [Background] Batalla A, Janssen H, Gangadin SS, Bossong MG. The Potential of Cannabidiol as a Treatment for Psychosis and Addiction: Who Benefits Most? A Systematic Review. J Clin Med. 2019 Jul 19;8(7):1058. doi: 10.3390/jcm8071058. PMID 31330972
- [Background] Hurd YL, Yoon M, Manini AF, Hernandez S, Olmedo R, Ostman M, Jutras-Aswad D. Early Phase in the Development of Cannabidiol as a Treatment for Addiction: Opioid Relapse Takes Initial Center Stage. Neurotherapeutics. 2015 Oct;12(4):807-15. doi: 10.1007/s13311-015-0373-7. PMID 26269227
- [Background] Paulus V, Billieux J, Benyamina A, Karila L. Cannabidiol in the context of substance use disorder treatment: A systematic review. Addict Behav. 2022 Sep;132:107360. doi: 10.1016/j.addbeh.2022.107360. Epub 2022 May 7. PMID 35580370